CLINICAL TRIAL: NCT06214039
Title: Virtual Reality Based Cognitive Behavioral Therapy for Public Speaking Anxiety
Brief Title: Virtual Reality Exposure for Public Speaking Anxiety
Acronym: VRanx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Linkoeping University (Other Government); Stockholm University (Other); Thomas More University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRanx_001
Record Dates: First submitted 2023-12-18; First posted 2024-01-19 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-11

CONDITIONS: Public Speaking Anxiety
Keywords: public speaking anxiety; virtual reality; social anxiety; psychological intervention; exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One session therapy (Active Comparator): One session exposure therapy followed by 4 weeks of internet-delivered self-help with therapist support on demand
  Interventions: Behavioral: Exposure in virtual reality and text based cognitive behavioral therapy (CBT) for public speaking anxiety
- One session therapy - divided into 3 (Experimental): Three session exposure therapy followed by 4 weeks of internet-delivered self-help with therapist support on demand
  Interventions: Behavioral: Exposure in virtual reality and text based cognitive behavioral therapy (CBT) for public speaking anxiety

INTERVENTIONS:
Behavioral: Exposure in virtual reality and text based cognitive behavioral therapy (CBT) for public speaking anxiety — A 3-hour one session exposure therapy for public speaking anxiety

SUMMARY:
This study aims to examine the efficacy of exposure using virtual reality (VR) for public speaking anxiety in young adults in two treatment arms: a one-session VR exposure therapy with a 4-week online transition intervention versus a three-session VR exposure therapy with a 4-week online transition intervention. Previous studies have demonstrated that one-session therapy (OST) is comparable to prolonged exposure-based therapies in terms of effectively reducing public speaking anxiety. Moreover, VR offers many benefits compared to in-person exposure, namely the ability to produce anxiety-evoking stimuli without having to leave the therapist's room. However, OST VR exposure has not been directly compared to prolonged VR exposure and not for public speaking anxiety.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30 and studying in higher education;
* experiencing a significant level of public speaking anxiety (60+ on PSAS);
* able to use a computer and have access to the internet for the duration of the study;
* able to understand, write and speak in Lithuanian;
* available to participate in one or three in-person intervention sessions and can devote the time to participate in a 4-week online program following the intervention sessions.

Exclusion Criteria:

* a history of seizures or a history of epilepsy;
* other significant medical conditions that would prevent them from participating in the program;
* high levels of depression (Patient Health Questionnaire-9 rating of 15 and above and mentions of suicidal ideation) or other significant psychiatric conditions that would interfere with participation in the program;
* a tendency to have extreme seasickness reactions or a history of adverse physical reactions to virtual reality experiences or difficulty with or lack of stereoscopic vision;
* current involvement in other psychological interventions such as psychological counseling or psychotherapy;
* use of psychoactive drugs, unless stable for three months;
* current participation in other programs aimed at reducing public speaking anxiety.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Public Speaking Anxiety Scale (PSAS), (Bartholomay & Houlihan, 2016). | Pre-treatment, mid-treatment, immediately after the intervention, 3 and 12 months post-treatment
  Canonical total score will be used. Measure is self-rated, online. The scale consists of 17 self-report statements measured on a Likert-type scale ranging from 1 "not at all", to 5 "extremely". A higher score indicates higher levels of experienced public speaking anxiety.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale - Self-Report (LSAS-SR), (Liebowitz, 2003; Rytwinski et al., 2009) | Pre-treatment, mid-treatment, immediately after the intervention, 3 and 12 months post-treatment
  Canonical total score will be used. Measure is self-rated, online. Items are rated using 4-point Likert scales ranging from 0 to 3. A higher score indicates more severe symptoms.
Brief Fear of Negative Evaluation Scale (BFNE), (Leary, 1983) | Pre-treatment, mid-treatment, immediately after the intervention, 3 and 12 months post-treatment
  Canonical total score will be used. Measure is self-rated, online. The BFNE is a 12-item, 5-point Likert-type scale, ranging from 1 ""not at all" to 5 "extremely". Higher scores indicate higher fear.
Igroup Presence Questionnaire (IPQ) | Pre-treatment, mid-treatment, immediately after the intervention, 3 and 12 months post-treatment
  Canonical total score will be used. Measure is self-rated, online. Each of the 14 items is rated on a 7-point Likert scale and the score is calculated by summing the ratings for each item.
Patient health questionnaire - 9 (PHQ-9), (Spitzer et al., 1999) | Pre-treatment, mid-treatment, immediately after the intervention, 3 and 12 months post-treatment
  Canonical total score will be used. Measure is self-rated, online. PHQ-9 consists of 9 items that are rated depending on how often the symptoms were bothersome using a 4-point scale, ranging from 0 "not at all" to 3 "nearly every day". The ratings are summed for the total score and higher scores indicates more severe depression symtpoms.

OTHER OUTCOMES:
Subjective Units of Distress (SUD) | Pre-intervention, immediately after the intervention
  Each measure will be rated on a scale from 0 to 100. Higher number indicates higher distress.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Eimontas, PhD, Study Chair — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Following the publication of trial results, participant-level data without identifying information, i.e., anonymized, will be stored on a national data archive MIDAS and will be made available to researchers affiliated with research institutions upon a reasonable request. Statistical analysis procedures will be clearly defined in papers on trial results.
Supporting Information: Study Protocol, SAP
Time Frame: Following the publication of the trial results.
Access Criteria: Available to researchers affiliated with research institutions upon a reasonable request.
URL: https://www.midas.lt